CLINICAL TRIAL: NCT02178436
Title: Phase Ib Study of the Selective Inhibitor of Nuclear Export (SINE) Selinexor (KPT-330), Gemcitabine and Nab-Paclitaxel and Phase II Study of Gemcitabine and Selinexor in Patients With Metastatic Pancreatic Cancer
Brief Title: Gemcitabine, Nab-paclitaxel and KPT-330 in Advanced Pancreatic Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mohammed Najeeb Al Hallak (Other)
Responsible Party: Sponsor-Investigator, Mohammed Najeeb Al Hallak, Principal Investigator, Barbara Ann Karmanos Cancer Institute
Organization: Barbara Ann Karmanos Cancer Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013-133; NCI-2014-01249 (Other: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2014-06-23; First posted 2014-06-30 (Estimated); Results first posted 2023-11-07 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: Acinar Cell Adenocarcinoma of the Pancreas; Duct Cell Adenocarcinoma of the Pancreas; Stage IV Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Gemcitabine; selinexor; Taxes; Albumin-Bound Paclitaxel

STUDY DESIGN:
Intervention Model Description: Phase I is completed, due to Dose Limiting Toxicities (DLT).
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Group I: Phase Ib (gemcitabine, nab-paclitaxel, selinexor) (Experimental): Patients receive gemcitabine hydrochloride IV, nab-paclitaxel IV, and selinexor PO on days 1, 8, and 15. Cycles repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: gemcitabine hydrochloride; Drug: Selinexor; Other: Pharmacological Study; Other: Laboratory Biomarker Analysis; Drug: Nab paclitaxel
- Group II: Phase II Group I (gemcitabine, selinexor) (Experimental): Patients receive gemcitabine hydrochloride IV on days 1, 8, and 15. Patients also receive selinexor PO on days 3, 8, and 15 of cycle 1 and on days 1, 8, and 15 for the subsequent cycles. Cycles repeat every 4 weeks in the absence of disease progression or unacceptable toxicity
  Interventions: Drug: gemcitabine hydrochloride; Drug: Selinexor; Other: Pharmacological Study; Other: Laboratory Biomarker Analysis
- GroupIII: Phase II Group II (gemcitabine, selinexor) (Experimental): Patients receive gemcitabine hydrochloride IV and selinexor PO on days 1, 8, and 15. Cycles repeat every 4 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: gemcitabine hydrochloride; Drug: Selinexor; Other: Pharmacological Study; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: gemcitabine hydrochloride — Given IV
  Other Names: dFdC; difluorodeoxycytidine hydrochloride; Gemcitabine HCI; Gemzar
Drug: Selinexor — Given IV
  Other Names: KPT-330; Xpovio; CRM1 nuclear export inhibitor KPT-330; selective inhibitor of nuclear export KPT-330; SINE KPT-330
Other: Pharmacological Study — Correlative studies
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Nab paclitaxel — Given IV
  Other Names: ABI 007; Abraxane; Protein-bound Paclitaxel; Nanoparticle Paclitaxel,
  Arms: Group I: Phase Ib (gemcitabine, nab-paclitaxel, selinexor)

SUMMARY:
This partially randomized phase Ib/II trial studies the side effects and best dose of selinexor when given together with gemcitabine and nab-paclitaxel, and to see how well they work in treating patients with pancreatic cancer that has spread to other parts of the body (metastatic). Drugs used in chemotherapy, such as selinexor, gemcitabine and nab-paclitaxel, work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading.

DETAILED DESCRIPTION:
Primary Objectives:

1. Phase I: To determine the recommended phase 2 dose (RP2D) of gemcitabine, nabpaclitaxel and selinexor for untreated metastatic pancreatic cancer [COMPLETED]
2. Phase I: To determine the safety profile of gemcitabine, nab-paclitaxel and selinexor [COMPLETED]
3. Phase II: To test whether the combination of gemcitabine and selinexor improves the median overall survival of patients with metastatic pancreatic cancer who have failed frontline non-gemcitabine containing regimens beyond 5.6 months (median overall survival of patient receiving gemcitabine only based on historical data.

Secondary Objectives:

1. To determine objective response rate to the combination of gemcitabine and selinexor using Response Evaluation Criteria in Solid Tumors (RECIST) criteria.
2. To assess safety of selinexor in combination with gemcitabine in phase II portion of the study
3. To determine progression free survival (PFS) in patients treated with gemcitabine and selinexor
4. To determine the influence of selinexor and gemcitabine on the nuclear expression and localization of tumor suppressor gene proteins.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent in accordance with federal, local, and institutional guidelines
* Patients with metastatic pancreatic adenocarcinoma not treated with chemotherapy for metastatic disease
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Absolute neutrophil count (ANC) >= 1500/mm^3
* Platelet count >= 100,000/mm^3
* Bilirubin < 2 times the upper limit of normal (ULN) (except patients with Gilbert's syndrome who must have a total bilirubin of < 3 times ULN)
* Alanine aminotransferase (ALT) < 2.5 times ULN
* Serum creatinine =< 1.5 mg/dL
* Serum albumin >= 3.0 g/dL
* Female patients of child-bearing potential must agree to use dual methods of contraception and have a negative serum pregnancy test at screening, and male patients must use an effective barrier method of contraception if sexually active with a female of child-bearing potential; acceptable methods of contraception are condoms with contraceptive foam, oral, implantable or injectable contraceptives, contraceptive patch, intrauterine device, diaphragm with spermicidal gel, or a sexual partner who is surgically sterilized or post-menopausal; for both male and female patients, effective methods of contraception must be used throughout the study and for three months following the last dose
* Patients with history of previously treated malignancies who have no evidence of disease for last five years are allowed to participate

Exclusion Criteria:

* Patients who are pregnant or lactating
* Radiation, chemotherapy, or immunotherapy or any other anticancer therapy =< 3 weeks prior to cycle 1 day 1; mitomycin C or radio-immunotherapy 6 weeks prior to cycle 1 day 1
* Major surgery within four weeks before cycle 1 day 1
* Unstable cardiovascular function:

  * Symptomatic ischemia, or
  * Uncontrolled clinically significant conduction abnormalities (e.g.: ventricular tachycardia on antiarrhythmics are excluded and 1st degree atrioventricular [AV] block or asymptomatic left anterior fascicular block [LAFB]/right bundle branch block [RBBB] will not be excluded), or
  * Congestive heart failure (CHF) of New York Heart Association (NYHA) class >= 3, or
  * Myocardial infarction (MI) within 3 months of cycle 1 day 1 dose
* Uncontrolled active infection requiring parenteral antibiotics, antivirals, or antifungals within one week prior to first dose
* Known to be HIV seropositive who are on anti-HIV drugs because of the unknown interactions between these drugs and the study agents
* Known active hepatitis A, B, or C infection; or known to be positive for hepatitis C virus (HCV) ribonucleic acid (RNA) or HBsAg (hepatitis B virus [HBV] surface antigen)
* Patients with active central nervous system (CNS) malignancy; asymptomatic small lesions are not considered active; treated lesions may be considered inactive if they are stable for at least 3 months
* Patients with significantly diseased or obstructed gastrointestinal tract or uncontrolled vomiting or diarrhea
* Grade >= 2 peripheral neuropathy within 14 days prior to cycle 1 day 1
* History of seizures, movement disorders or cerebrovascular accident within the past 5 years prior to cycle 1 day 1
* Patients with muscular degeneration, uncontrolled glaucoma, or markedly decreased visual acuity based on physician's assessment
* Serious psychiatric or medical conditions that could interfere with treatment
* Participation in an investigational anti-cancer study within 3 weeks prior to cycle 1 day 1
* Concurrent therapy with approved or investigational anticancer therapeutic
* Presence of clinically significant ascites

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2014-10-31 (Actual); Primary Completion 2021-11-27 (Actual); Study Completion 2023-04-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mohammed N Al Hallak, M.D., Principal Investigator — Barbara Ann Karmanos Cancer Institute
Locations (2):
- United States (2):
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Stony Brook University Cancer Center, Stony Brook, New York

REFERENCES:
- [Derived] Azmi AS, Khan HY, Muqbil I, Aboukameel A, Neggers JE, Daelemans D, Mahipal A, Dyson G, Kamgar M, Al-Hallak MN, Tesfaye A, Kim S, Shidham V, M Mohammad R, Philip PA. Preclinical Assessment with Clinical Validation of Selinexor with Gemcitabine and Nab-Paclitaxel for the Treatment of Pancreatic Ductal Adenocarcinoma. Clin Cancer Res. 2020 Mar 15;26(6):1338-1348. doi: 10.1158/1078-0432.CCR-19-1728. Epub 2019 Dec 12. PMID 31831564

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Accrual time period: 10/31/14 - 02/09/22
Pre-assignment Details: 2 patients enrolled but did not receive any treatment
Period: Overall Study
Arm/Group | Group I: Phase Ib (Gemcitabine, Nab-paclitaxel, Selinexor) | Group II: Phase II Group I (Gemcitabine, Selinexor) | GroupIII: Phase II Group II (Gemcitabine, Selinexor)
Started | 9 | 0 | 4
Completed | 9 | 0 | 4
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Group II enrolled no patients because patients refused to undergo the required biopsy.
Groups:
- Total: Total of all reporting groups
Arm/Group | Group I: Phase Ib (Gemcitabine, Nab-paclitaxel, Selinexor) | Group II: Phase II Group I (Gemcitabine, Selinexor) | GroupIII: Phase II Group II (Gemcitabine, Selinexor) | Total
Number analyzed (Participants) | 9 | 0 | 4 | 13
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 68 [61 to 73] |  | 56 [53 to 56.5] | 61 [56 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 |  | 2 | 6
  Male | 5 |  | 2 | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 |  | 0 | 0
  Not Hispanic or Latino | 8 |  | 3 | 11
  Unknown or Not Reported | 1 |  | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0 | 0
  Asian | 0 |  | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 |  | 0 | 0
  Black or African American | 2 |  | 1 | 3
  White | 6 |  | 2 | 8
  More than one race | 0 |  | 0 | 0
  Unknown or Not Reported | 1 |  | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 9 |  | 4 | 13

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD) of Selinexor, Gemcitabine Hydrochloride, and Paclitaxel Albumin-stabilized Nanoparticle Formulation Combination (Phase Ib)
Description: MTD is defined as the lowest dose for which less than a third of patients experience a dose limiting toxicity graded according to National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 4.03.
Time Frame: 28 days
Population: Maximum tolerated dose is only estimated using the Phase 1b samples
Measure: Number; unit: milligrams
Arm/Group | Group I: Phase Ib (Gemcitabine, Nab-paclitaxel, Selinexor) | Group II: Phase II Group I (Gemcitabine, Selinexor) | GroupIII: Phase II Group II (Gemcitabine, Selinexor)
Number analyzed (Participants) | 9 | 0 | 0
milligrams | 80 |  |

2. Primary Outcome: Proportion of Patients With a Toxic Event, Graded According to NCI CTCAE Version 4.03
Description: The reported output is the proportion of patients that had a toxic event along with the associated 90% Wilson's confidence interval.
Time Frame: Up to 2 years
Population: Group II enrolled no patients because patients refused to undergo the required biopsy.
Measure: Number (90% Confidence Interval); unit: proportion of patients
Arm/Group | Group I: Phase Ib (Gemcitabine, Nab-paclitaxel, Selinexor) | Group II: Phase II Group I (Gemcitabine, Selinexor) | GroupIII: Phase II Group II (Gemcitabine, Selinexor)
Number analyzed (Participants) | 9 | 0 | 4
proportion of patients | 1.00 [0.77 to 1.00] |  | 0.75 [0.36 to 0.94]

3. Primary Outcome: Overall Survival (Phase II)
Description: Estimated on an intention-to-treat basis (using all registered patients), and on a response-evaluable basis (using all patients who completed at least one 4-week treatment cycle) using the Kaplan-Meier method.
Time Frame: Up to 7 months post treatment initiation
Population: Group II enrolled no patients because patients refused to undergo the required biopsy.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Group I: Phase Ib (Gemcitabine, Nab-paclitaxel, Selinexor) | Group II: Phase II Group I (Gemcitabine, Selinexor) | GroupIII: Phase II Group II (Gemcitabine, Selinexor)
Number analyzed (Participants) | 9 | 0 | 4
months | 5.45 [4.37 to NA] — Median survival (MS) is calculated by using the Kaplan-Meier (KM) curve. The MS is found by seeing where the estimated KM curve intersects with the horizontal line indicating 50% survival (HL-50). The upper 90% confidence value for the MS is found by seeing where the upper confidence band (CB) for the KM estimate intersects with HL-50. For this analysis, the upper CB does not cross 0.5 for the whole time period under study; so it never intersects with HL-50; and thus is not available to report |  | NA [NA to NA] — No survival events occurred in this group during the follow-up time. Therefore a median survival and confidence interval are not estimable.

4. Secondary Outcome: Effects the Study Drug Combination Has on Participants
Description: Pharmacodynamics of selinexor in combination with gemcitabine hydrochloride and paclitaxel albumin-stabilized nanoparticle formulation
Time Frame: Day 1 of course 1 (before selinexor administration, 1, 2, 4 and 8 hours after selinexor administration) and days 2, 3 and 8
Population: Pharmacodynamics data was not measured.
Arm/Group | Group I: Phase Ib (Gemcitabine, Nab-paclitaxel, Selinexor) | Group II: Phase II Group I (Gemcitabine, Selinexor) | GroupIII: Phase II Group II (Gemcitabine, Selinexor)
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Proportion of Patients With a Response
Description: Point and 90% Wilson's confidence intervals will be estimated to describe response rate. If the best observed clinical response was complete response or partial response, we consider that the patient responded.
Time Frame: Up to 2 years
Population: Group II enrolled no patients because patients refused to undergo the required biopsy. Four patients in Group I were not evaluated for response.
Measure: Number (90% Confidence Interval); unit: proportion of patients
Arm/Group | Group I: Phase Ib (Gemcitabine, Nab-paclitaxel, Selinexor) | Group II: Phase II Group I (Gemcitabine, Selinexor) | GroupIII: Phase II Group II (Gemcitabine, Selinexor)
Number analyzed (Participants) | 5 | 0 | 4
proportion of patients | 0.40 [0.14 to 0.73] |  | 0 [0 to 0.40]

6. Secondary Outcome: Progression Free Survival (Phase II)
Description: Estimated on an intention-to-treat basis (using all registered patients), and on a response-evaluable basis (using all patients who completed at least one 4-week treatment cycle) using the Kaplan-Meier method. Both progression and death are considered events for this analysis.
Time Frame: Up to 2 years
Population: Group II enrolled no patients because patients refused to undergo the required biopsy.
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Group I: Phase Ib (Gemcitabine, Nab-paclitaxel, Selinexor) | Group II: Phase II Group I (Gemcitabine, Selinexor) | GroupIII: Phase II Group II (Gemcitabine, Selinexor)
Number analyzed (Participants) | 9 | 0 | 4
months | 4.60 [4.37 to NA] — Median survival (MS) is calculated by using the Kaplan-Meier (KM) curve. The MS is found by seeing where the estimated KM curve intersects with the horizontal line indicating 50% survival (HL-50). The upper 90% confidence value for the MS is found by seeing where the upper confidence band (CB) for the KM estimate intersects with HL-50. For this analysis, the upper CB does not cross 0.5 for the whole time period under study; so it never intersects with HL-50; and thus is not available to report |  | 1.74 [1.22 to NA] — Median survival (MS) is calculated by using the Kaplan-Meier (KM) curve. The MS is found by seeing where the estimated KM curve intersects with the horizontal line indicating 50% survival (HL-50). The upper 90% confidence value for the MS is found by seeing where the upper confidence band (CB) for the KM estimate intersects with HL-50. For this analysis, the upper CB does not cross 0.5 for the whole time period under study; so it never intersects with HL-50; and thus is not available to report

7. Other Pre Specified Outcome: Change in Gene Expression (Including Forkhead Box Protein O, I-kappaB, Cyclin-dependent Kinase Inhibitor 1B, Par4 and Phosphorylated Signal Transducer and Activator of Transcription 3) (Phase II)
Description: Seven patients in each group will yield a two-sided 90% confidence interval with a distance from the mean change to the limits of 0.75 standard deviation units. A two-sided p-value of 0.10 will be used for all analyses.
Time Frame: Baseline to up to 2 years
Population: Gene expression data was not measured.
Arm/Group | Group I: Phase Ib (Gemcitabine, Nab-paclitaxel, Selinexor) | Group II: Phase II Group I (Gemcitabine, Selinexor) | GroupIII: Phase II Group II (Gemcitabine, Selinexor)
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: The adverse events were collected from cycle one day one of study treatment until four weeks follow up visit or thirty days after study treatment was discontinued up to 2 years.
Description: No patients were enrolled in Group 2, so the number of patients at risk is 0 for that group.
Arm/Group | Group I: Phase Ib (Gemcitabine, Nab-paclitaxel, Selinexor) | Group II: Phase II Group I (Gemcitabine, Selinexor) | GroupIII: Phase II Group II (Gemcitabine, Selinexor)
All-Cause Mortality (participants affected / at risk) | 9/9 | 0/0 | 0/4
Serious Adverse Events (participants affected / at risk) | 6/9 | 0/0 | 0/4
Other Adverse Events (participants affected / at risk) | 9/9 | 0/0 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group I: Phase Ib (Gemcitabine, Nab-paclitaxel, Selinexor) (N=9) | Group II: Phase II Group I (Gemcitabine, Selinexor) (N=0) | GroupIII: Phase II Group II (Gemcitabine, Selinexor) (N=4)
Abdominal Pain (Gastrointestinal disorders) | 1 | 0 | 0
Cognitive disturbance (Nervous system disorders) | 1 | 0 | 0
Death NOS (General disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0
Hyperglycemia (Investigations) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0
Psychiatric disorders - Other (Psychiatric disorders) | 1 | 0 | 0
Renal and urinary disorders - Other (Renal and urinary disorders) | 1 | 0 | 0
Stroke (Nervous system disorders) | 1 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 1 | 0 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group I: Phase Ib (Gemcitabine, Nab-paclitaxel, Selinexor) (N=9) | Group II: Phase II Group I (Gemcitabine, Selinexor) (N=0) | GroupIII: Phase II Group II (Gemcitabine, Selinexor) (N=4)
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0
Alanine aminotransferase increased (Investigations) | 2 | 0 | 0
Alkaline phosphatase increased (Investigations) | 1 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 0 | 0
Anemia (Blood and lymphatic system disorders) | 1 | 0 | 1
Anorexia (Gastrointestinal disorders) | 4 | 0 | 0
Anxiety (Psychiatric disorders) | 2 | 0 | 0
Ascites (Gastrointestinal disorders) | 1 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 0
Blood bilirubin increased (Investigations) | 1 | 0 | 0
Blurred vision (Eye disorders) | 2 | 0 | 0
Bruising (Injury, poisoning and procedural complications) | 1 | 0 | 0
Chills (General disorders) | 2 | 0 | 0
Constipation (Gastrointestinal disorders) | 2 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Creatinine increased (Investigations) | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 3 | 0 | 0
Depression (Psychiatric disorders) | 2 | 0 | 0
Diarrhea (Gastrointestinal disorders) | 7 | 0 | 1
Dizziness (Nervous system disorders) | 2 | 0 | 1
Dry mouth (Gastrointestinal disorders) | 1 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 6 | 0 | 0
Dysgeusia (Nervous system disorders) | 4 | 0 | 0
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 1 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1
Eye disorders - Other, specify (Eye disorders) | 4 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 3 | 0 | 0
Fatigue (General disorders) | 8 | 0 | 0
Flashing lights (Eye disorders) | 1 | 0 | 0
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 | 0 | 0
General disorders and administration site conditions - Other, specify (General disorders) | 1 | 0 | 0
Headache (Nervous system disorders) | 1 | 0 | 0
Hemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0
Hot flashes (Vascular disorders) | 1 | 0 | 0
Hyperglycemia (Investigations) | 1 | 0 | 0
Hypoalbuminemia (Investigations) | 1 | 0 | 0
Hypoglycemia (Investigations) | 1 | 0 | 0
Hypokalemia (Investigations) | 1 | 0 | 1
Infections and infestations - Other, specify (Infections and infestations) | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 1 | 0 | 0
Malaise (General disorders) | 3 | 0 | 0
Mucositis oral (Gastrointestinal disorders) | 1 | 0 | 0
Musculoskeletal and connective tissue disorder - Other, specify (Metabolism and nutrition disorders) | 2 | 0 | 0
Nausea (Gastrointestinal disorders) | 8 | 0 | 0
Neuralgia (Nervous system disorders) | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 3 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 5 | 0 | 0
Platelet count decreased (Blood and lymphatic system disorders) | 1 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Psychiatric disorders - Other, specify (Psychiatric disorders) | 1 | 0 | 0
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin infection (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Upper respiratory infection (Infections and infestations) | 1 | 0 | 0
Urinary frequency (Renal and urinary disorders) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 7 | 0 | 0
Weight loss (Investigations) | 1 | 0 | 1
White blood cell decreased (Blood and lymphatic system disorders) | 2 | 0 | 0
Edema limbs (General disorders) | 3 | 0 | 0
Oral dysesthesia (Nervous system disorders) | 1 | 0 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1 | 0 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 1
Hyponatremia (Investigations) | 0 | 0 | 1
Rectal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-18): https://cdn.clinicaltrials.gov/large-docs/36/NCT02178436/Prot_SAP_000.pdf